CLINICAL TRIAL: NCT04350788
Title: Enhancing Survivorship Care Planning for Patients With Localized Prostate Cancer Using A Couple-focused Web-based Tailored Symptom Self-management Program
Acronym: SCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LCCC 1619; 1R21CA212516 (NIH)
Record Dates: First submitted 2020-03-28; First posted 2020-04-17 (Actual); Results first posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: survivorship care plan; quality of life; supportive care
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Survivorship Care Plan (SCP) (Placebo Comparator): The SCP group (control) participants were directed to the National Cancer Institute PC website (NCI) (http://www.cancer.gov/types/prostate),
  Interventions: Other: Survivorship Care Plan
- Enhanced SCP (ESCP) (Experimental): ESCP consists of the standard SCP that is enhanced by a couple-focused, tailored mHealth PC education program, the Patient Education Resources for Couples, to improve symptom management at home.
  Interventions: Other: Enhanced Survivorship Care Plan

INTERVENTIONS:
Other: Survivorship Care Plan — Participants visit the NCI prostate cancer website in addition to their standardized post-treatment survivorship care
  Arms: Survivorship Care Plan (SCP)
Other: Enhanced Survivorship Care Plan — In addition to their standardized post-treatment survivorship care, participants visit the prostate cancer education resources for couples (PERC) website that was based on scientific evidence and input from stakeholders including PC patients, partners, and cancer care providers. Participants learn about skills and knowledge about how to enhance their positive appraisals of symptoms and self-efficacy in symptom management through information and skills training, fostering healthy behaviors, and facilitating social support
  Arms: Enhanced SCP (ESCP)

SUMMARY:
The purpose of this research study is to examine the feasibility of the enhanced survivorship care plans (ESCPs, regular SCPs with the a web-based couple-focused symptom self-management project (PERC) or National Cancer Institute prostate cancer web links) and to conduct an initial benefit assessment of enhanced survivorship care plans among prostate cancer patients transitioning from active treatment to post-treatment self-management, and their partners.

Participation of this study lasts for about for 16 weeks. Depending on participants' need for information, it takes 10-30 minutes of their time each week to review the information about prostate cancer.

Eligible and consented patients with newly treated localized prostate cancer and your partner (couples) are randomly assigned to the regular survivorship care plan (SCPs) with the NCI website or the enhanced survivorship care plans (SCP plus the web-based prostate cancer education program, PERC) groups. They complete baseline (T1, prior to randomization) and 4-month post-T1 follow-up measures (T2).

DETAILED DESCRIPTION:
Methods: A two-group randomized controlled pretest-posttest design will be used and collect data at baseline (T1) and 4 months later (T2) among 50 patients completing initial treatment for localized prostate cancer and their partners. First, the investigators will assess the feasibility of ESCP by recruitment, enrollment, and retention rates, program satisfaction with the ESCP, and perceived ease of use of the ESCP. To achieve the secondary aim, the ESCP users will be compared with the standardized SCP users and assess their primary outcomes of QOL (overall, physical, emotional, and social QOL), secondary outcomes (reduction in negative appraisals and improvement in self-efficacy, social support, and health behaviors to manage symptoms), and number of visits to post-treatment care services at T1 and T2. The primary and secondary outcomes are assessed using measurements with sound psychometrical properties. The investigators will use a qualitative and quantitative mixed methods approach to achieve the research aims.

Conclusions: The results from this study will help design a definitive randomized trial to test the efficacy of the ESCPs, a potentially scalable program, to enhance supportive care for prostate cancer patients and their families.

ELIGIBILITY:
Inclusion Criteria:

Eligibility included men who:

* were diagnosed with localized PC;
* were within 16 weeks of completing their initial curative intent treatment [26] at genitourinary and radiation oncology clinics at two comprehensive cancer centers in the U.S southeast;
* were not treated for another cancer in last year; and
* had a partner > 18 years of age not receiving cancer treatment.

Exclusion Criteria:

* Either member of couple unable to speak English
* Unwilling/unable to provide Informed Consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Song, RN, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months following publication
Access Criteria: Investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Song L, Guo P, Tan X, Chen RC, Nielsen ME, Birken SA, Koontz BF, Northouse LL, Mayer DK. Enhancing survivorship care planning for patients with localized prostate cancer using a couple-focused web-based, mHealth program: the results of a pilot feasibility study. J Cancer Surviv. 2021 Feb;15(1):99-108. doi: 10.1007/s11764-020-00914-7. Epub 2020 Jul 17. PMID 32681304

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: dyad
Period: Overall Study
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
Started | 62; 31 dyad | 62; 31 dyad
Completed | 50; 25 dyad | 56; 28 dyad
Not Completed | 12; 6 dyad | 6; 3 dyad
Not completed — Lost to Follow-up | 6 | 2
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Protocol Violation | 4 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: dyad
Groups:
- Total: Total of all reporting groups
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP) | Total
Number analyzed (Participants) | 62 | 62 | 124
Number analyzed (dyad) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.63 (7.37) | 62.62 (8.13) | 63.12 (7.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 31 | 31 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 46 | 44 | 90
  Black | 13 | 16 | 29
  Other | 3 | 2 | 5
Education [Count of Participants; unit: Participants]
  Less than college | 28 | 29 | 57
  Bachelor's Degree | 17 | 14 | 31
  Graduate Degree (Master's PhD, JD, MD, etc.) | 17 | 19 | 36
Employment Status [Count of Participants; unit: Participants]
  Yes | 32 | 34 | 66
  No | 30 | 28 | 58
Income [Count of Participants; unit: Participants] — the range of household's current annual income
  Participants
    <= $60,000 | 20 | 17 | 37
    >$60,000 | 34 | 39 | 73
    Don't know/refused | 8 | 6 | 14
Type of Treatment [Count of Units; unit: dyad]
  Radiation | 16 | 17 | 33
  Surgery | 15 | 14 | 29
Charlson comorbidity index [Mean (Standard Deviation); unit: score on a scale] — Charlson comorbidity index is a weighted scale of comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis codes. The index range is (0,19). Lower score indicates less severe comorbid condition.
  score on a scale | 3.85 (1.76) | 4.21 (2.18) | 4.03 (1.98)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Potentially Eligible Participants Actually Enrolled Into the Study
Description: Will evaluate the percentage of patients and partners successfully consented and completing the baseline survey among all people approached for the study
Time Frame: after participants completed baseline survey
Population: We excluded 62 of the 211 patients who we approached but did not meet the eligibility criteria. For 149 patients who met study criteria, we asked if they were willing to participant the study. We contacted partners only if patients consented.
Measure: Count of Units; unit: dyad
Units Other Than Participants: dyad
Groups:
- Overall: Enrollment rate is calculated before randomization without arms.
Arm/Group | Overall
Number analyzed (Participants) | 149
Number analyzed (dyad) | 149
dyad | 62

2. Primary Outcome: Percentage of Participants Enrolled Who Remained in the Study and Completed the Post-Intervention Follow-Up Survey
Description: Will evaluate the percentage of participants successfully following protocol, defined as completing the Follow-Up survey at the end of the study period among those who have been enrolled into the study (who completed the baseline).
Time Frame: during 4-month study period
Measure: Count of Units; unit: dyad
Units Other Than Participants: dyad
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
Number analyzed (Participants) | 62 | 62
Number analyzed (dyad) | 31 | 31
dyad | 25 | 28

3. Primary Outcome: Percentage of Participants That Used the Web-Based Intervention Sessions That Are Consistent With Patient-Reported Symptoms
Description: The usage of Web-Based Intervention Sessions is determined by the percentage of participants who logged into the study website among those who have been randomly assigned to the intervention group. Patient-Reported Symptoms are determined by patient's responses on their appraisal of prostate cancer symptoms and general symptoms. 1=patient reported the symptom and the symptom webpage reviewed; 0=patient reported the symptom and no related webpage reviewed OR patient did not report the symptom but the webpage reviewed
Time Frame: during 4-month study period
Population: We don't have information about web pages that participants reviewed in control group.
Measure: Count of Units; unit: dyad
Units Other Than Participants: dyad
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
Number analyzed (Participants) | 0 | 62
Number analyzed (dyad) | 0 | 31
dyad |  | 13

4. Primary Outcome: Participant Satisfaction Scores
Description: Program satisfaction determined by the 11-item Participant Satisfaction Scale measured the level of program satisfaction. The first to tenth items ranged from 1=not satisfied to 5=extremely satisfied. The eleventh item ranged from 1=extremely not to 4=definitely yes. Higher total score indicates greater program satisfaction
Time Frame: at the 4 month followup
Population: Intention-to-treat was used in analyses. The sample size was 124 participants (62 patient-partner couples in each group) who completed baseline and were randomized. We analyzed group differences by role (patient vs partner).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Survivorship Care Plan (SCP): Patient; Survivorship Care Plan (SCP): Partner: The SCP group (control) participants were directed to the National Cancer Institute PC website (NCI) (http://www.cancer.gov/types/prostate),
  Survivorship Care Plan: Participants visit the NCI prostate cancer website in addition to their standardized post-treatment survivorship care
- Enhanced SCP (ESCP): Patient; Enhanced SCP (ESCP): Partner: ESCP consists of the standard SCP that is enhanced by a couple-focused, tailored mHealth PC education program, the Patient Education Resources for Couples, to improve symptom management at home.
  Enhanced Survivorship Care Plan: In addition to their standardized post-treatment survivorship care, participants visit the prostate cancer education resources for couples (PERC) website that was based on scientific evidence and input from stakeholders including PC patients, partners, and cancer care providers. Participants learn about skills and knowledge about how to enhance their positive appraisals of symptoms and self-efficacy in symptom management through information and skills training, fostering healthy behaviors, and facilitating social support
Arm/Group | Survivorship Care Plan (SCP): Patient | Enhanced SCP (ESCP): Patient | Survivorship Care Plan (SCP): Partner | Enhanced SCP (ESCP): Partner
Number analyzed (Participants) | 31 | 31 | 31 | 31
score on a scale | 30.48 (11.47) | 36.30 (8.11) | 36.29 (13.54) | 38.59 (10.34)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP): Patient vs Enhanced SCP (ESCP): Patient; We analyzed program satisfaction between SCP and ESCP by role (patient vs partner). The following result is for patient; Test type: Superiority; p = 0.02, t-test, 1 sided
Statistical Analysis 2: Comparison: Survivorship Care Plan (SCP): Patient vs Enhanced SCP (ESCP): Patient; We analyzed program satisfaction between SCP and ESCP by role (patient vs partner). The following result is for partner; Test type: Superiority; p = 0.25, t-test, 1 sided

5. Primary Outcome: Perceived Ease of Use Score
Description: The 16-item Program Usability measures participants' assessment of their agreement with the ease of use of the program in terms of its general features, content, and navigation. The ranges of the total scores are (3,15), (4,20), (9,45) for general features, content, and navigation, respectively. The score of individual item ranges from1=strongly disagree to 5=strongly agree. Higher score indicates greater perceived ease of use.
Time Frame: at the 4 month followup
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survivorship Care Plan (SCP): Patient | Enhanced SCP (ESCP): Patient | Survivorship Care Plan (SCP): Partner | Enhanced SCP (ESCP): Partner
Number analyzed (Participants) | 31 | 31 | 31 | 31
score on a scale
  General | 12.44 (1.58) | 12.60 (1.29) | 12.68 (1.53) | 12.53 (1.58)
  Content | 17.11 (2.37) | 17.32 (1.99) | 16.83 (2.26) | 16.55 (2.21)
  Navigation | 33.89 (5.26) | 36.84 (3.93) | 34.79 (4.80) | 35.02 (5.66)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP): Patient vs Enhanced SCP (ESCP): Patient; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for patient in general domain; Test type: Superiority; p = 0.36, t-test, 1 sided
Statistical Analysis 2: Comparison: Survivorship Care Plan (SCP): Patient vs Enhanced SCP (ESCP): Patient; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for patient in content domain; Test type: Superiority; p = 0.38, t-test, 1 sided
Statistical Analysis 3: Comparison: Survivorship Care Plan (SCP): Patient vs Enhanced SCP (ESCP): Patient; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for patient in navigation domain; Test type: Superiority; p = 0.02, t-test, 1 sided
Statistical Analysis 4: Comparison: Survivorship Care Plan (SCP): Partner vs Enhanced SCP (ESCP): Partner; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for partner in general domain; Test type: Superiority; p = 0.62, t-test, 1 sided
Statistical Analysis 5: Comparison: Survivorship Care Plan (SCP): Partner vs Enhanced SCP (ESCP): Partner; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for partner in content domain; Test type: Superiority; p = 0.65, t-test, 1 sided
Statistical Analysis 6: Comparison: Survivorship Care Plan (SCP): Partner vs Enhanced SCP (ESCP): Partner; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for partner in navigation domain; Test type: Superiority; p = 0.45, t-test, 1 sided

6. Secondary Outcome: Change in FACT-G Scores
Description: Change in QOL determined using the Functional Assessment of Cancer Therapy General Scale (FACT-G) v.4, a 27-item measure yielding total score and scores for physical, social/family, emotional, and functional well-being of demonstrated reliability, validity, and sensitivity to change. FACT-G consists of 4 subscales: physical well-being (PWB), functional well-being (FWB), emotional well-being (EWB) and social well-being (SWB). Scores on the four subscales are summed to produce a total score ranging from 0 to 108 with higher scores indicating better quality of life. Change from baseline is the post-Baseline values minus the Baseline value.
Time Frame: Baseline upon enrollment, Month 4
Population: Intention-to-treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
Number analyzed (Participants) | 62 | 62
score on a scale | -0.03 (8.98) | 1.91 (8.38)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP) vs Enhanced SCP (ESCP); Test type: Superiority; p = 0.35, Mixed Models Analysis

7. Secondary Outcome: Change in Appraisal of Prostate Cancer-Specific Symptoms
Description: The Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. EPIC will be used to measure change in appraisal of symptoms scores among patients from Baseline (T1) to T2 (4 months post T1). EPIC contains 26 items within 5 domains: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing opposite results by role: patient with better appraisal of symptoms and partner with worse appraisal of symptoms. Change from baseline is the post-Baseline values minus the Baseline value.
Time Frame: Baseline upon enrollment, Month 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survivorship Care Plan (SCP): Patient | Enhanced SCP (ESCP): Patient | Survivorship Care Plan (SCP): Partner | Enhanced SCP (ESCP): Partner
Number analyzed (Participants) | 31 | 31 | 31 | 31
score on a scale
  Urinary | 11.03 (16.91) | 19.58 (23.02) | -0.48 (0.87) | -0.46 (1.75)
  Bowel | 2.31 (8.83) | 6.93 (20.17) | -0.2 (1.00) | -0.11 (1.10)
  Sexual | 1.46 (21.01) | 7.45 (22.54) | 0.04 (1.40) | 0.32 (1.31)
  Hormonal | 1.99 (17.48) | 4.61 (15.81) | -0.04 (1.21) | -0.21 (1.47)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP): Patient vs Enhanced SCP (ESCP): Patient; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for patient in urinary domain; Test type: Superiority; p = 0.01, ANCOVA
Statistical Analysis 2: Comparison: Survivorship Care Plan (SCP): Patient vs Enhanced SCP (ESCP): Patient; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for patient in bowel domain; Test type: Superiority; p = 0.41, ANCOVA
Statistical Analysis 3: Comparison: Survivorship Care Plan (SCP): Patient vs Enhanced SCP (ESCP): Patient; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for patient in sexual domain; Test type: Superiority; p = 0.21, ANCOVA
Statistical Analysis 4: Comparison: Survivorship Care Plan (SCP): Patient vs Enhanced SCP (ESCP): Patient; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for patient in hormonal domain; Test type: Superiority; p = 0.52, ANCOVA
Statistical Analysis 5: Comparison: Survivorship Care Plan (SCP): Partner vs Enhanced SCP (ESCP): Partner; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for partner in urinary domain; Test type: Superiority; p = 0.79, ANCOVA
Statistical Analysis 6: Comparison: Survivorship Care Plan (SCP): Partner vs Enhanced SCP (ESCP): Partner; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for partner in bowel domain; Test type: Superiority; p = 0.84, ANCOVA
Statistical Analysis 7: Comparison: Survivorship Care Plan (SCP): Partner vs Enhanced SCP (ESCP): Partner; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for partner in sexual domain; Test type: Superiority; p = 0.82, ANCOVA
Statistical Analysis 8: Comparison: Survivorship Care Plan (SCP): Partner vs Enhanced SCP (ESCP): Partner; We analyzed this measure between SCP and ESCP by role (patient vs partner) and by domain. The following result is for partner in hormonal domain; Test type: Superiority; p = 0.33, ANCOVA

8. Secondary Outcome: Change in Appraisal of General Symptoms
Description: The 19-item Risk for Distress-general symptoms is a subscale of the Risk for Distress Scale. It measures how much trouble the participant has with the general symptoms such as pain, fatigue, and etc. The total score ranges between 0 and 38, with higher scores indicating worse appraisal of symptoms. Change from baseline is the post-Baseline values minus the Baseline value.
Time Frame: Baseline upon enrollment, Month 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survivorship Care Plan (SCP): Patient | Enhanced SCP (ESCP): Patient | Survivorship Care Plan (SCP): Partner | Enhanced SCP (ESCP): Partner
Number analyzed (Participants) | 31 | 31 | 31 | 31
score on a scale | -1.26 (4.21) | -2.97 (5.26) | -0.59 (4.26) | -1.35 (4.27)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP): Patient vs Enhanced SCP (ESCP): Patient; Test type: Superiority; p = 0.18, ANCOVA
Statistical Analysis 2: Comparison: Survivorship Care Plan (SCP): Partner vs Enhanced SCP (ESCP): Partner; Test type: Superiority; p = 0.38, ANCOVA

9. Secondary Outcome: Healthcare Utilization Extracted From Electronic Medical Record
Description: The total number of prostate cancer-related followup visits, emergency room use and readmissions.
Time Frame: during the first 10 months after participants completed baseline survey
Population: Intention-to-treat was used in analyses. The overall number of participants analyzed was 62 patients (62 patient-partner couples in each group) who completed baseline and were randomized. Because we would like to analyze the intervention effects on patient's healthcare utilization.
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
Number analyzed (Participants) | 31 | 31
number of visits | 4.84 (4.68) | 4.65 (4.56)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP) vs Enhanced SCP (ESCP); Test type: Superiority; p = 0.05, generalized linear regression

10. Secondary Outcome: Change in Self-Efficacy Scores From Baseline to 4-Months Post Baseline
Description: The Lewis Cancer Self-Efficacy used to measure change in participants' feelings of self-efficacy in dealing with the patient's cancer diagnosis and treatment from Baseline (T1) to T2 (4 months post T1). Participants rate statements about how confident they feel on a scale from 1 to 10, where higher scores indicate higher self-efficacy.
Time Frame: Baseline upon enrollment, Month 4
Population: Intention-to-treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
Number analyzed (Participants) | 62 | 62
score on a scale | -1.40 (6.81) | 0.50 (5.58)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP) vs Enhanced SCP (ESCP); Test type: Superiority; p = 0.10, Mixed Models Analysis

11. Secondary Outcome: Change in PROMIS Social Support-Informational Support From Baseline to 4-Months Post-Baseline
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Informational Support Short Form 8a will be used to assess changes in patient and partner reported informational support system using a 5-point Likert scale from Baseline (T1) to T2 (4 months post T1). The total score range: 8-40. Higher scores indicate more informational support. Change from baseline is the post-Baseline values minus the Baseline value.
Time Frame: Baseline upon enrollment, Month 4
Population: Intention-to-treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
Number analyzed (Participants) | 62 | 62
score on a scale | -0.09 (8.81) | 0.98 (6.24)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP) vs Enhanced SCP (ESCP); Test type: Superiority; p = 0.29, Mixed Models Analysis

12. Secondary Outcome: Change in PROMIS Social Support-Emotional Support From Baseline to 4-months Post-Baseline
Description: The PROMIS Emotional Support System-Short Form 8a will be used to assess changes in the self-reported emotional support system of patients and their partners using a 5-point Likert scale from Baseline (T1) to T2 (4 months post T1). The total score range: 8-40. Higher scores indicate more emotional social support. Change from baseline is the post-Baseline values minus the Baseline value.
Time Frame: Baseline upon enrollment, Month 4
Population: Intention-to-treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
Number analyzed (Participants) | 62 | 62
score on a scale | 0.02 (6.74) | 0.29 (5.93)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP) vs Enhanced SCP (ESCP); Test type: Superiority; p = 0.49, Mixed Models Analysis

13. Secondary Outcome: Change in PROMIS Social Support-Instrumental Support From Baseline to 4-months Post-Baseline
Description: The PROMIS Instrumental Support-Short Form 8a will be used to assess changes in patient and partner reported instrumental support system using a 5-point Likert scale from Baseline (T1) to T2 (4 months post T1). The total score range: 8-40. Higher scores indicate more instrumental support. Change from baseline is the post-Baseline values minus the Baseline value.
Time Frame: Baseline upon enrollment, Month 4
Population: Intention-to-treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
Number analyzed (Participants) | 62 | 62
score on a scale | -0.76 (6.59) | -0.21 (5.76)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP) vs Enhanced SCP (ESCP); Test type: Superiority; p = 0.09, Mixed Models Analysis

14. Secondary Outcome: Change in Dietary Risk Assessment Scores From Baseline to 4-month Post Baseline as Measured by the Health Promoting Lifestyle Profile II
Description: Change in Dietary Risk Assessment scores used to measure changes in dietary risk from Baseline (T1) to T2 (4 months post T1). Change from baseline is the post-Baseline values minus the Baseline value. Participants are asked how often they consume different foods over the past month or week and respond using a Likert Scale ranging from 1=never to 4=routinely. The total score range: 8-32. Higher scores indicate better health behaviors in nutrition.
Time Frame: Baseline upon enrollment, Month 4
Population: Intention-to-treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
Number analyzed (Participants) | 62 | 62
score on a scale | -0.10 (0.43) | -0.10 (0.44)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP) vs Enhanced SCP (ESCP); Test type: Superiority; p = 0.16, Mixed Models Analysis

15. Secondary Outcome: Change in Physical Activity Assessment Scores From Baseline to 4-month Post Baseline as Measured by the Health Promoting Lifestyle Profile II
Description: Change in Physical Activity Assessment scores used to measure changes in physical activity from Baseline (T1) to T2 (4 months post T1). Change from baseline is the post-Baseline values minus the Baseline value. Participants are asked how often they engage in exercises and physical activity over the past month or week and respond using a Likert Scale, ranging from 1=never to 4=routinely. The total score range: 9-36. Higher scores indicate better health behaviors in physical activity.
Time Frame: Baseline upon enrollment, Month 4
Population: Intention-to-treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
Number analyzed (Participants) | 62 | 62
score on a scale | -0.02 (0.51) | -0.01 (0.49)
Statistical Analysis 1: Comparison: Survivorship Care Plan (SCP) vs Enhanced SCP (ESCP); Test type: Superiority; p = 0.55, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 2 years from the beginning of the study recruitment to the end of data collection.
Description: No death happened during the study period, and thus, the All-Cause Mortality is zero
Arm/Group | Survivorship Care Plan (SCP) | Enhanced SCP (ESCP)
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 2/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Survivorship Care Plan (SCP) (N=62) | Enhanced SCP (ESCP) (N=62)
restarting cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — After consent and enrollment, it was discovered that the patient started another round of radiation treatment during the study, making both the patient and his partner ineligible for our dyadic study. There is only one event.
Severe health problem (Cardiac disorders) | 0 (0) | 1 (1) — The patient was hospitalized for about two months after having a stroke, and thus, made both the patient and his partner ineligible in the study. This is however only one event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT04350788/Prot_SAP_000.pdf